CLINICAL TRIAL: NCT00556439
Title: Concurrent Pilot Studies in Giant Cell Arteritis and Takayasu's Arteritis to Examine the Safety, Efficacy, and Immunologic Effects of Abatacept (CTLA4-Ig) in Large Vessel Vasculitis
Brief Title: Abatacept for Treating Adults With Giant Cell Arteritis and Takayasu's Arteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: The Cleveland Clinic (Other); Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR070018; 268200700036C-5-0-1 (NIH); HHSN2682007000036C; NCT00788268 (obsolete NCT alias)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Takayasu's Arteritis; Giant Cell Arteritis
Keywords: Vasculitis; Arteritis; Takayasu's; Temporal Arteritis; Abatacept
MeSH Terms: conditions — Takayasu Arteritis; Giant Cell Arteritis; Vasculitis; Arteritis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A and C (Experimental): This is a randomized withdrawal design protocol. All participants will receive abatacept and prednisone (a glucocorticoid) for the first 3 months. Abatacept will be given intravenously on selected days. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Month 3, and finally further tapered until discontinuation is reached. At Month 3, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to abatacept at this point will be in Group A for giant cell arteritis and Group C for Takayasu arteritis.
  Interventions: Drug: Abatacept
- B and D (Placebo Comparator): This is a randomized withdrawal design protocol. All participants will receive abatacept and prednisone (a glucocorticoid) for the first 3 months. Abatacept will be given intravenously on selected days. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Month 3, and finally further tapered until discontinuation is reached. At Month 3, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to placebo at this point will be in Group B for giant cell arteritis and Group D for Takayasu arteritis.
  Interventions: Drug: Abatacept; Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Participants will receive a fixed dose of abatacept, approximating 10mg per kilogram of body weight. The following dosing rules will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  Abatacept will be administered in a 30-minute intravenous infusion on Days 1, 15, 29 (Month 1) and at Month 2. In the absence of toxicity or relapse, participants will remain on abatacept at the same dosage until randomization at Month 3. After randomization, only Group A (giant cell arteritis) and Group C (Takayasu arteritis) participants will continue on abatacept.
  Other Names: Orencia
Drug: Placebo — Placebo abatacept infusions will be given monthly after random assignment at Month 3.
  Arms: B and D

SUMMARY:
Giant cell arteritis (GCA) and Takayasu's arteritis (TAK) are diseases that cause swelling of the arteries in the head, neck, upper body, and arms. TAK specifically affects the aorta, the largest blood vessel in the body, and its branches. Therapies are available to improve the symptoms of GCA and TAK, but relapse often occurs, and better treatments are needed. Abatacept is a drug that interacts with certain cells in the body that are involved with GCA and TAK. This study will evaluate the effectiveness of abatacept in treating GCA and TAK and preventing disease relapse.

DETAILED DESCRIPTION:
GCA and TAK both cause inflammation in the lining of the arteries, which can interfere with the body's ability to carry oxygen to areas that need it. Symptoms of GCA include headaches, jaw pain, and blurred or double vision. Serious symptoms that occur less commonly are blindness and stroke. TAK symptoms include fever, fatigue, weight loss, arthritis, and non-specific aches and pains. There may also be tenderness near affected arteries. Researchers believe that GCA and TAK are diseases that are controlled by the body's immune system. Activated T-cells, specifically, are critical to the origin and development of these diseases. Abatacept is a medication that modulates the signal required for T-cell activation. This study will evaluate the safety and effectiveness of abatacept in treating GCA and TAK and preventing disease relapse.

Participation in this study may last up to 4 years. Participants will receive abatacept intravenously on specified days during Months 1, 2, and 3. They will also receive daily prednisone, which will be started at a dose of 40 to 60mg, then tapered to 20mg by Month 3, and finally further tapered until discontinuation is reached. At Month 3, participants who have achieved remission will be randomly assigned under double-blind conditions to either continue abatacept or be switched to placebo infusions. Both treatments will be given once a month at study visits. Blood samples will also be collected at the monthly study visits to conduct laboratory-based studies. Participants who remain in remission will continue to receive abatacept or placebo monthly until the common closing date, defined as 12 months after enrollment of the 33rd participant for each disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GCA or TAK (defined below)
* History of active GCA or TAK within the past 2 months
* Age of 15 years or older
* Willing to use an effective means of birth control throughout the study

Specific Inclusion Criteria for Participants with GCA:

* Participants must meet three of the following five criteria, including either Criterion 4 or 5:

  1. Age at disease onset was equal to or greater than 50 years
  2. Disease onset was recent or experiencing a new type of localized pain in the head
  3. Erythrocyte sedimentation rate greater than 40mm in the first hour, as determined using the Westergren method
  4. Temporal artery abnormality (i.e., temporal artery tenderness to palpation or decreased pulsation, unrelated to arteriosclerosis of cervical arteries)
  5. Temporal artery or large vessel biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cell or characteristic changes of large vessel stenosis or aneurysm by arteriography

Specific Inclusion Criteria for Participants with TAK:

* Presence of abnormalities that are consistent with TAK identified using arteriography, plus at least one of the following criteria:

  1. Age at disease onset was less than 50 years
  2. Pain in the legs or arms
  3. Decreased brachial artery pulse (one or both arteries)
  4. Difference of more than 10mm Hg in blood pressure between the arms
  5. Bruit over subclavian arteries or aorta

Exclusion Criteria:

* Evidence of active infection (including chronic infection)
* Pregnant or breastfeeding
* HIV infected, hepatitis C infected, or a positive hepatitis B surface antigen
* Inability to comply with study guidelines
* Inability to provide informed consent
* Cytopenia, as defined by a platelet count of less than 80,000/mm3, an absolute neutrophil count of less than 1,500/mm3, and hematocrit less than 20%
* Insufficient kidney function, as defined by a serum creatinine of more than 3 mg/dL or creatinine clearance of 20 ml/min or less
* Other uncontrolled disease that could prevent safe study completion
* History of any malignant neoplasm except adequately treated basal or squamous cell carcinoma of the skin or solid tumors treated with curative therapy and disease-free for at least 5 years
* Receipt of an investigational agent or device within 30 days prior to study entry
* A live vaccination within 4 weeks prior to study entry
* Presence of a positive tuberculin skin test with induration of at least 5mm
* Radiographic evidence suggestive of tuberculosis
* Poor tolerability of blood draws or lack of adequate access to veins for medication administration and blood draws
* History of treatment with rituximab within 12 months prior to study entry or history of treatment with rituximab more than 12 months prior to study entry, where the B lymphocyte count has not returned to normal
* History of treatment with infliximab within the past 49 days, adalimumab within the past 28 days, or etanercept within the past 21 days.
* Presence of any of the following diseases or conditions:

  1. Microscopic polyangiitis
  2. Churg-Strauss syndrome
  3. Polyarteritis nodosa
  4. Cogan's syndrome
  5. Behcet disease
  6. Sarcoidosis
  7. Kawasaki disease
  8. Tuberculosis or atypical mycobacterial infection
  9. Deep fungal infection
  10. Lymphoma, lymphomatoid granulomatosis, or other type of malignancy that mimics vasculitis
  11. Cryoglobulinemic vasculitis
  12. Systemic lupus erythematosus
  13. Rheumatoid arthritis
  14. Mixed connective tissue disease or any overlap autoimmune syndrome

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Langford, MD, MHS, Principal Investigator — The Cleveland Clinic
Locations (10):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Hospital, Hamilton, Ontario
  - Mt. Sinai Hospital Toronto, Toronto, Ontario

REFERENCES:
- [Derived] Langford CA, Cuthbertson D, Ytterberg SR, Khalidi N, Monach PA, Carette S, Seo P, Moreland LW, Weisman M, Koening CL, Sreih AG, Spiera R, McAlear CA, Warrington KJ, Pagnoux C, McKinnon K, Forbess LJ, Hoffman GS, Borchin R, Krischer JP, Merkel PA; Vasculitis Clinical Research Consortium. A Randomized, Double-Blind Trial of Abatacept (CTLA-4Ig) for the Treatment of Takayasu Arteritis. Arthritis Rheumatol. 2017 Apr;69(4):846-853. doi: 10.1002/art.40037. Epub 2017 Mar 8. PMID 28133931
- [Derived] Langford CA, Cuthbertson D, Ytterberg SR, Khalidi N, Monach PA, Carette S, Seo P, Moreland LW, Weisman M, Koening CL, Sreih AG, Spiera R, McAlear CA, Warrington KJ, Pagnoux C, McKinnon K, Forbess LJ, Hoffman GS, Borchin R, Krischer JP, Merkel PA; Vasculitis Clinical Research Consortium. A Randomized, Double-Blind Trial of Abatacept (CTLA-4Ig) for the Treatment of Giant Cell Arteritis. Arthritis Rheumatol. 2017 Apr;69(4):837-845. doi: 10.1002/art.40044. Epub 2017 Mar 3. PMID 28133925
- [Derived] Goldstein BL, Gedmintas L, Todd DJ. Drug-associated polymyalgia rheumatica/giant cell arteritis occurring in two patients after treatment with ipilimumab, an antagonist of ctla-4. Arthritis Rheumatol. 2014 Mar;66(3):768-9. doi: 10.1002/art.38282. No abstract available. PMID 24574239
- See also: Click here for the Cleveland Clinic Center for Vasculitis Care and Research Web site — http://www.clevelandclinic.org/arthritis/vasculitis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with giant cell arteritis or Takayasu arteritis were recruited at 11 academic medical centers. For giant cell arteritis, the first participant was enrolled 2/2009 and the last participant was enrolled 1/2014. For Takayasu arteritis, the first participant was enrolled 2/2009 and the last participant was enrolled 11/2013.
Groups:
- Group A - Abatacept in Giant Cell Arteritis: This is a randomized withdrawal design protocol. Participants with giant cell arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to abatacept at this point will be in Group A.
- Group B - Placebo in Giant Cell Arteritis: This is a randomized withdrawal design protocol. All participants with giant cell arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to placebo at this point will be in Group B.
- Group C - Abatacept in Takayasu Arteritis: This is a randomized withdrawal design protocol. Participants with Takayasu arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to abatacept at this point will be in Group C.
- Group D - Placebo in Takayasu Arteritis: This is a randomized withdrawal design protocol. All participants with Takayasu arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to placebo at this point will be in Group D.
Period: Study Entry to Week 12
Arm/Group | Group A - Abatacept in Giant Cell Arteritis | Group B - Placebo in Giant Cell Arteritis | Group C - Abatacept in Takayasu Arteritis | Group D - Placebo in Takayasu Arteritis
Started | 49 (58 signed informed consent with 9 not being eligible. The remaining 49 received study drug.) | 0 (No participants received placebo until the Week 12 Randomization) | 34 (39 signed informed consent with 5 not being eligible. The remaining 34 received study drug.) | 0 (No participants received placebo until the Week 12 Randomization)
Completed | 41 | 0 | 26 | 0
Not Completed | 8 | 0 | 8 | 0
Not completed — Lack of Efficacy | 5 | 0 | 6 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Recurrent infection | 1 | 0 | 0 | 0
Not completed — Malignancy | 0 | 0 | 1 | 0
Period: After Week 12 (Randomized Study Period)
Arm/Group | Group A - Abatacept in Giant Cell Arteritis | Group B - Placebo in Giant Cell Arteritis | Group C - Abatacept in Takayasu Arteritis | Group D - Placebo in Takayasu Arteritis
Started | 20 | 21 | 11 | 15
Completed | 17 | 17 | 11 | 14
Not Completed | 3 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Malignancy | 0 | 1 | 0 | 1
Not completed — Severe infection | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Reflects the population that reached Week 12 blinded randomization. In the giant cell arteritis cohort, 8 of 49 were withdrawn at or before Week 12 with a total of 41 remaining in the active comparator group. In the Takayasu arteritis cohort, 8 of 34 were withdrawn at or before Week 12 with a total of 26 remaining in the active comparator group.
Groups:
- Group A - Abatacept in Giant Cell Arteritis: This is a randomized withdrawal design protocol. All participants with giant cell arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to abatacept at this point will be in Group A.
- Group C - Abatacept in Takayasu Arteritis: This is a randomized withdrawal design protocol. All participants with Takayasu arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to abatacept at this point will be in Group C.
- Total: Total of all reporting groups
Arm/Group | Group A - Abatacept in Giant Cell Arteritis | Group B - Placebo in Giant Cell Arteritis | Group C - Abatacept in Takayasu Arteritis | Group D - Placebo in Takayasu Arteritis | Total
Number analyzed (Participants) | 20 | 21 | 11 | 15 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 11 | 15 | 40
  >=65 years | 9 | 18 | 0 | 0 | 27
Age, Continuous [Median (Full Range); unit: Years] | 63.47 [57.27 to 80.13] | 71.48 [54.26 to 86.63] | 30.17 [18.93 to 58.94] | 28.61 [19.54 to 56.97] | 48.74 [19.93 to 86.63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 9 | 13 | 59
  Male | 4 | 0 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 21 | 10 | 14 | 62
  Unknown or Not Reported | 3 | 0 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 19 | 19 | 8 | 12 | 58
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 5 | 3 | 3 | 17
  United States | 14 | 16 | 8 | 12 | 50

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome - Relapse-free Survival (RFS)
Description: Relapse: presence of active disease occurring after a period of remission
  Remission: absence of active disease
  Active disease defined by clinical features or imaging or both:
  Clinical features:
  1 or more of the following attributed to GCA/TAK:
  * Sustained fever of >38 C for > 1 week
  * Vascular pain/tenderness > 1 day, non-fleeting
  * Headache a) present > 1 day b) non-fleeting c) not relieved with analgesics d) not typical for pre-existing headaches
  * Ischemic retinopathy, optic neuropathy, or visual loss
  * Tongue/jaw pain and/or claudication
  * TIA or stroke
  * Extremity claudication
  * Musculoskeletal symptoms + ESR of > 40 mm/hr or CRP above the normal limit
  * Malaise/fatigue + ESR of > 40 mm/hr or CRP above the normal limit
  * Other symptoms/signs due to GCA/TAK requiring reinstitution/increase in GC
  Imaging features
  • Development of new vascular stenosis or aneurysm in new vascular territories as seen by MRI/MRA or arteriogram
Time Frame: Weeks 0 to 64
Population: The primary study endpoint was relapse-free survival (RFS). Kaplan-Meier curves of RFS were constructed for each stratum (giant cell arteritis and Takayasu arteritis), and differences in treatment arms compared using the logrank test. The analysis of the primary outcome was based upon intent to treat.
Measure: Count of Participants; unit: Participants
Groups:
- Group D - Placebo in Takayasu Arteritis: This is a randomized withdrawal design protocol. Participants with Takayasu arteritis will receive prednisone (a glucocorticoid) and abatacept for the first 12 weeks. Prednisone will be started at a dose of 40 to 60mg, then tapered to 20mg by Week 12 and finally further tapered until discontinuation is reached at Week 28. Abatacept will be given intravenously on Day 1, Day 15, and Week 8 at a fixed dose approximating 10mg per kilogram of body weight. The following dosing rules for abatacept will be followed:
  * Participants weighing less than 60kg will receive 500mg of abatacept.
  * Participants weighing 60 to 100kg will receive 750mg of abatacept.
  * Participants weighing more than 100kg will receive 1000mg of abatacept.
  At Week 12, participants who have achieved remission will be randomly assigned under double-blind conditions to receive monthly infusions of either abatacept or placebo. Participants who are assigned to placebo at this point will be in Group D.
Arm/Group | Group A - Abatacept in Giant Cell Arteritis | Group B - Placebo in Giant Cell Arteritis | Group C - Abatacept in Takayasu Arteritis | Group D - Placebo in Takayasu Arteritis
Number analyzed (Participants) | 20 | 21 | 11 | 15
Participants
  Relapsed | 10 | 14 | 8 | 10
  Remained in remission | 10 | 7 | 3 | 5
Statistical Analysis 1: Comparison: Group A - Abatacept in Giant Cell Arteritis vs Group B - Placebo in Giant Cell Arteritis; The planned sample size was determined by the minimally clinically meaningful result (i.e., an approximate 30% improvement in relapse-free survival) to be detected utilizing a one-sided alpha of 0.1. Kaplan-Meier curves of RFS were constructed for each stratum, and differences in treatment arms compared using the logrank test. The analysis of the primary outcome was based upon intent to treat; Test type: Other — Kaplan-Meier curves of relapse free survival were constructed, and differences in treatment arms compared using the logrank test. The analysis of the primary outcome was based upon intent to treat; p = 0.049, Log Rank — The p value of 0.049 reflects comparison of relapse free survival of abatacept versus placebo in giant cell arteritis
Statistical Analysis 2: Comparison: Group C - Abatacept in Takayasu Arteritis vs Group D - Placebo in Takayasu Arteritis; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.853, Log Rank — The p value of 0.853 reflects comparison of relapse free survival of abatacept versus placebo in Takayasu arteritis

ADVERSE EVENTS:
Time Frame: Week 0 to end of study
Description: Toxicity grades were assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE). Expected or unexpected adverse events that were grade 1 were not collected or reported.
Arm/Group | Group A - Abatacept in Giant Cell Arteritis | Group B - Placebo in Giant Cell Arteritis | Group C - Abatacept in Takayasu Arteritis | Group D - Placebo in Takayasu Arteritis
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 8/20 | 5/21 | 5/11 | 7/15
Other Adverse Events (participants affected / at risk) | 14/20 | 15/21 | 8/11 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Abatacept in Giant Cell Arteritis (N=20) | Group B - Placebo in Giant Cell Arteritis (N=21) | Group C - Abatacept in Takayasu Arteritis (N=11) | Group D - Placebo in Takayasu Arteritis (N=15)
Ocular/visual - other (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Branch retinal artery occlusion - 1 event, Transient vision loss - presumed due to GCA - 1 event
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative-injury - other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Total knee replacement
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Post-operative deep venous thrombosis
Gastrointestinal - other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Diarrhea/dehydration
Dermatology /Skin - other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Herpes zoster - 1 event - abatacept, Squamous cell carcinoma - 1 event - placebo
Metabolic/laboratory - other (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hyperglycemia
Infection with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Diverticulitis
Bone: spine-scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Spinal surgery
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Syncope
Pain - other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Narcotic withdrawal
Pulmonary/Upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Dyspnea - 1 event, COPD - 1 event
Renal/genitourinary - other (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Endometrial carcinoma - 1 event Transitional cell carcinoma - 1 event
Urinary electrolyte wasting (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Urine electrolyte disturbance
Gastrointestinal - other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Ischemic colitis
Ulcer - GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Duodenal ulcer
Hemorrhage - GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Ischemic colitis - 1 event, Rectal bleeding - 1 event
Infection - other (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Possible pyelonephritis - 1 event - abatacept, Skin site infection post thrombectomy - 1 event - abatacept, Pyelonephritis - 1 event - placebo, Epiglottitis - 1 event - placebo
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Appendicitis - 1 event, Nausea/vomiting/diarrhea due to possible infection - 1 event
Pain - other (General disorders) | 0 (0) | 0 (0) | 2 (7) | 1 (1) — Non cardiac chest pain - 6 events in 1 participant - abatacept, Headache due to Migraine - 1 event - abatacept, Chest pain unclear etiology - 1 event - placebo
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Dyspnea/dysphagia due to GERD
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Arterial thrombosis following angioplasty
Vascular - other (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Elective aortic surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Abatacept in Giant Cell Arteritis (N=20) | Group B - Placebo in Giant Cell Arteritis (N=21) | Group C - Abatacept in Takayasu Arteritis (N=11) | Group D - Placebo in Takayasu Arteritis (N=15)
Blood and bone marrow - other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrhythmia - other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatology - other (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endocrine - other (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroid (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - other (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - other (Infections and infestations) | 5 (10) | 7 (10) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
ALT, SGPT (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
AST, SGOT (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic/laboratory - other (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis non-septic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint - function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal/Soft tissue - other (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood alteration (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Ocular/Visual - other (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - other (General disorders) | 1 (4) | 1 (1) | 0 | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary - other (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hearing (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac general - other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Endocrine - other (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection - other (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 7 (17)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (9)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (6)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST, SGOT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Albumin, serum - low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calcium, serum - low (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose, serum - high (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Glucose, serum - low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Metabolic/laboratory - other (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sodium, serum - low (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurology - other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular/visual - other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain - other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular - other (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, challenges in assessing disease activity in giant cell arteritis and Takayasu arteritis, 84.6% of patients with Takayasu arteritis were enrolled for the treatment of a disease relapse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No